CLINICAL TRIAL: NCT05548803
Title: Comparing Patient-reported Impact of COVID-19 Shelter-in-place Policies and Access to Containment and Mitigation Strategies, Overall and in Vulnerable Populations
Brief Title: COVID-19 Citizen Science Expansion Project
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Sutter Health (Other); Carelon Research (Other); Louisiana Public Health Institute (Other); Duke University (Other); New York University (Other); Albert Einstein College of Medicine (Other); University of Utah (Other); Ochsner Health System (Other); Baylor Scott and White Health (Other); Wake Forest University Health Sciences (Other); New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 20203090
Record Dates: First submitted 2022-09-19; First posted 2022-09-21 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 Citizen Science (CCS), launched in March 2020, supports collaborative research on symptoms, risk factors, surveillance, biomarkers and testing for COVID-19 using the Eureka Research Platform. CCS maintains IRB approval with UCSF's IRB (UCSF IRB# 17-21879).

This CCS Expansion Project, which is funded jointly by the National Institutes of Health (NIH), the Patient-Centered Outcomes Research Institute (PCORI), and the Bill and Melinda Gates Foundation, will invite patients at health systems across the US to contribute their health records data and then join the established CCS study, allows for linked analysis of CCS data and health records data, and provides the scientific rationale and plan for the project.

DETAILED DESCRIPTION:
Shelter-in-place orders, social distancing, and mandatory closure of non-essential businesses across the country have suppressed transmission of SARS-CoV-2 and limited direct health impact of the COVID-19 Pandemic. These policies, however, exact an enormous societal cost and cannot be maintained indefinitely. When and how to lift restrictions represents the defining challenge of our time for local, state and national leaders, and requires excruciating decisions that balance lives lost from coronavirus infection against economic, social and indirect health effects of restrictive policy. To understand the impact of these decisions, we must hear from patients. We propose to recruit a large population-based sample of PCORnet patients into our digital cohort of "COVID-19 Citizen Scientists," gather patient-reported outcomes with linked electronic health record (EHR), and analyze it to answer the following critical research questions (RQs):

RQ1: What is the comparative impact of different shelter-in-place/reopening policies, overall and in vulnerable populations, on patient-reported financial insecurity, mental health, and other subjective outcomes important to patients? The natural experiment that occurs as state governors and local county health departments across the US differentially lift and/or reinstate shelter-in-place policies, and that is ongoing today as the US considers reopening fully (despite threats from new coronavirus variants), represents an analytic opportunity to estimate and compare benefits and harms of different policies, both overall and for vulnerable subsets of the population. To leverage this opportunity, we will collect a detailed record of county- (and state-) level COVID-19-related policies, including shelter-in-place (aka containment & closure), economic response and public health policies, starting at the beginning of the Pandemic in March 2020 and continuing through the end of the year into 2021. We have selected 119 counties for data collection where we have the most patient-reported survey responses through 2020, and where we expect to enroll many new participants through Fall 2021. We will use these data to analyze the impact on patient-reported outcomes, and then make them available to other investigators.

RQ2: What is the comparative effectiveness of county-level containment and mitigation strategies at achieving timely access to COVID-19 vaccination (overall and among previously hesitant persons), testing, healthcare, information, and contact tracing, overall and in vulnerable populations? Timely access to containment and mitigation strategies were (and will continue to be) critical to quickly detect and slow transmission of coronavirus and future pandemics in communities, and to effectively care for patients who become infected. Unlike shelter-in-place policies that are highly publicized, containment and mitigation strategies are about resource allocation and operational effectiveness. Decision-making may be hidden, but we can measure the effectiveness of these strategies by asking patients. For example, we can assess reasons for vaccination among participants that were previously hesitant, delays in coronavirus testing after patients develop symptoms using our daily symptom survey data to provide the denominator (all symptomatic patients) and the anchor time point (time of symptom onset); and weekly surveys will assess access to critical information (e.g., "Do you know how to get a COVID-19 test?") and contact tracing after testing positive.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Has the capacity to read and comprehend English
3. Has internet access and a device (computer, tablet, laptop, etc.) that can access it

Exclusion Criteria:

1. Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our goal will be to recruit a large sample of participants that is representative of the US population. In particular, we wish to make inferences about Hispanic/LatinX and African- American/Black subsets of the US population, who appear to be especially vulnerable to both direct (infection-related) and indirect impact of the Pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 54689 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
GAD-7 anxiety score | Over the course of the pandemic, up to 5 years
  Anxiety is measured in monthly surveys using the seven-item General Anxiety Disorder-7 (GAD-7) questionnaire. Responses to each item in the GAD-7 are scored as integer values between 0-3 according to the frequency of symptoms during the preceding two weeks ("Not at all", "Several days", "More than half the days", or "Nearly every day"). The sum of all seven items produces a combined score between 0-21, where scores ≥ 10 are considered indicative of moderate to severe anxiety disorders

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pletcher, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (9):
- United States (9):
  - Sutter Health, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Advocate Aurora Health, Downers Grove, Illinois
  - Ochsner Health System, New Orleans, Louisiana
  - NYC Health + Hospitals, New York, New York
  - New York University, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Baylor Scott and White Health, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No